CLINICAL TRIAL: NCT06688084
Title: Evaluation of Pathogenicity Factors of Staphylococcus Pettenkoferi in Foot Wounds and Osteitis in Diabetic Patients
Brief Title: Pathogenicity Factors of Staphylococcus Pettenkoferi in Foot Wounds and Osteitis in Diabetic Patients
Acronym: PETTENK-OS
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Staphylococcal National Reference Center, Lyon, France (Unknown); Rennes University Hospital (Other); Nantes University Hospital (Other); Universität Tübingen (Other); Örebro University, Sweden (Other); Charles University, Czech Republic (Other); University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2023-2/CM-01
Record Dates: First submitted 2024-11-09; First posted 2024-11-14 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes; Foot; Infection; Staphylococcus pettenkoferi; Osteitis
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Infections; Osteitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — This is an international multi-center translational research project, based on a collection of strains (strain library) consisting of 230 S. pettenkoferi isolates collected between 2015 and 2023 from 9 European centres, (Reference 2021U1047-002).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Molecular epidemiology of the collection — Next-generation genomic sequencing (MICRO&BIO platform, MiSeq, Illumina) and bioinformatics analyses. After validating data quality, genomes will be re-assembled using Spades software (version 3.15.4) and CLC® (Qiagen), then compared with the National Center for Biotechnology Information GenBank database. They will also be analysed on the online Type-Strain Genomes Server platform to accurately identify the bacteria. Genome annotation will be done using the DDBJ Fast Annotation and Submission Tool. Single nucleotide polymorphisms (SNP) analysis based on the alignment of whole genomes and core-genomes will be carried out using version 7 of MAFFT (multiple alignment using fast Fourier transform) software, then quantified using snp-dists (version 0.6.3). This approach will enable the molecular epidemiology of the collection of strains in France and other European countries to be clarified, and the main circulating clades to be assessed, particularly depending on the origin of samples.
Other: Study of the resistome of the S. pettenkoferi population — The resistome will be assessed by identifying known and described resistance genes in staphylococci using bioinformatics analyses of sequenced complete bacterial genomes. A search for plasmids will also be made using various specific software packages (ResFinder, CARD, PointFinder, Plasmidfinder, in-house pipeline).
Other: Study of the virulome of the S. pettenkoferi population — The virulome of the strains will be studied based on the genomic sequencing data obtained and with reference to the literature on Staphylococci. Various specific software packages (Pathogenfinder, Virulencefinder, in-house pipeline) will be used for this purpose.
Other: Study of the resistance profiles of all S. pettenkoferi isolates — Antibiotic resistance will be assessed using a Sensititer® plate (Thermo ScientificTM, Illkirch) to evaluate the minimum inhibitory concentration of isolates against a series of antibiotics commonly used for S. pettenkoferi infections, including new molecules currently on the market or in development, such as Ceftaroline, Ceftobiprole, Dalbavancin, Delafloxacin, Tedizolid and Oritavancin. Minimum inhibitory concentration values will be interpreted in accordance with the recommendations of the Antibiogram Committee of the Société Française de Microbiologie (https://www.sfm-microbiologie.org/2021/04/23/casfm-avril-2021-v1-0/).
Other: Selection of strains for in-depth phenotypic study — Different strains of S. pettenkoferi isolated from foot osteitis in diabetic patients and non-diabetic osteitis will be selected according to the clades identified and phenotypically characterised by further analysis:
  * Observation of culture characteristics (culture requirements, growth time, colony size and haemolytic capacity), (n=20)
  * Determination of growth curves by measuring absorbance at 600 nm using the Infinite M Mano automatic absorbance reader (TECAN, Lyon), (n=20)
  * Study of the ability to form biofilm in the presence (antibiofilmogram) (n=85) or absence (BioFilm Ring® test, Biofilm Control, St Beauzire) (n=85) of various antibiotics commonly used for the treatment of S. pettenkoferi infection during osteitis.
Other: Selection of strains (n=3) for the virulence study — Three strains of S. pettenkoferi isolated from foot osteitis in diabetic patients will be selected on the basis of the clades identified and the study of the virulome in order to be analysed on :
  * In vitro cell culture models of macrophages (RAW 264.7) and osteoblasts (MC3T3-E1) to assess the invasion potential of these isolates by measuring internalisation rates (TECAN, Lyon) and LDH release (CyQUANT LDH Cytotoxicity kit), a sign of cellular toxicity of the isolate.
  * An in vivo wound model on diabetic zebrafish (Dario rerio) with evaluation of their survival at 48h in the presence of the isolates by immersion.
  These models were developed at the MICRO&BIO Platform and the INSERM 1047 VBIC unit.

SUMMARY:
Gram-positive cocci, particularly Staphylococcus aureus and coagulase-negative staphylococci (SCoN), are the bacteria most frequently isolated from diabetic foot ulcers. Although studies have been carried out on the role of S. aureus in the unfavorable evolution of these wounds, no studies have focused on the role of SCoN. Of the fifty or so SCoN species, not all have the same virulence potential. The role of Staphylococcus pettenkoferi is unknown, yet this bacterium is the 7th most frequently identified in diabetic foot ulcers, suggesting that it may also be involved in the pathophysiology of these infections. At Nîmes University Hospital, this bacterium is mainly identified in samples from diabetic foot ulcers or osteitis in our laboratory and 80% of the bacteria present are in biofilms.It is essential to understand the mechanisms governing these bacterial interactions and establish the true pathogenic potential of these bacteria. Recently, the Nîmes team showed that a strain of S. pettenkoferi (SP165) isolated from foot osteitis in a diabetic patient had real virulence potential. SP165 could not only produce biofilm, but could also survive in human blood, human keratinocytes and murine and human macrophages. It also caused significant embryonic mortality in a zebrafish model. A second study of 29 isolates from Nîmes University Hospital subsequently demonstrated that there were two predominant clones with different virulences. Three biofilm production profiles (rapidly and highly biofilm-producing, slowly biofilm-producing and non-biofilm-producing) and two zebrafish profiles (highly and moderately lethal) were reported by phenotypic and genomic analyses on this panel of strains. Genes for resistance, virulence and biofilm production were also found on their genomes.

DETAILED DESCRIPTION:
Gram-positive cocci, in particular Staphylococcus aureus and coagulase-negative staphylococci (SCoN), are the bacteria most frequently isolated from diabetic foot ulcers. While studies have been carried out on the role of S. aureus in the unfavorable evolution of these wounds, no study has focused on the role of SCoN. Of the fifty or so SCoN species, not all have the same virulence potential. The role of Staphylococcus pettenkoferi is not known. Yet this bacterium is the 7th most frequently identified in diabetic foot ulcers, suggesting that it may also be involved in the pathophysiology of these infections. In the work of Loetsche et al. a study of the microbiome of 349 diabetic foot ulcer samples by targeted 16S rDNA sequencing showed that the genus Staphylococcus was the most abundant, with a relative abundance of 22.8%, including 13.3% S. aureus and 5.3% S. pettenkoferi.

At Nîmes University Hospital, this bacterium is mainly identified in samples from diabetic foot ulcers or osteitis in our laboratory (89 isolations of S. pettenkoferi from diabetic foot ulcer samples out of 167 isolations made of this bacterium between 2018 and 2022).The difficulty of managing chronic wounds also lies in the fact that almost 80% of the bacteria present are in biofilms. It has also been established that the environment in which bacteria are found, and in particular the interactions they establish between themselves, play a significant role in delayed wound healing. It is therefore essential to understand the mechanisms governing these bacterial interactions and to establish the true pathogenic potential of these bacteria.

Recently, our team demonstrated that a strain of S. pettenkoferi (SP165) isolated from foot osteitis in a diabetic patient had real virulence potential. As well as being able to produce biofilm, SP165 was able to survive in human blood, human keratinocytes and murine and human macrophages. It also demonstrated its virulence by causing significant embryonic mortality in the zebrafish model.

A second study of 29 isolates from Nîmes University Hospital subsequently demonstrated the existence of two predominant clones with different virulences.

Three biofilm production profiles (rapidly and highly biofilm-producing, slowly biofilm-producing and non-biofilm-producing) and two zebrafish virulence profiles (highly and moderately lethal) were reported by phenotypic and genomic analyses on this panel of strains. Genes for resistance, virulence and biofilm production were also found on their genomes.

ELIGIBILITY:
Inclusion Criteria:

* Not applicable for this research on a ready-constituted collection of strains of Staphylococcus pettenkoferi

Exclusion Criteria:

* Not applicable for this research on a ready-constituted collection of strains of Staphylococcus pettenkoferi

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The collection of strains at the Nîmes University Hospital site from 9 European laboratories collected between 2015 and 2023 for a total of 108 months was carried out between November 2021 and August 2023.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Genetic diversity of Staphyloccocus pettenkoferi strains isolated from osteitis and non-diabetic wounds, blood cultures and nasal carriage. | Day 0 to 3 months
  Number of clades estimated via typing by complete sequencing of the bacterial genomes of all S. pettenkoferi strains and analysis of phylogenetic distances (whole genome and core genome single nucleotide polymorphisms).

SECONDARY OUTCOMES:
Genetic diversity of Staphyloccocus pettenkoferi strains isolated from osteitis and non-diabetic wounds, blood cultures and nasal carriage. | 3 - 6 months
  Number of clades estimated via typing by complete sequencing of the bacterial genomes of all Staphylococcus pettenkoferi strains and analysis of phylogenetic distances.
Resistome in the strain population according to sample origin:osteitis | 3 - 6 months
  The presence of antibiotic resistance genes (resistome) will be identified by bioinformatics analysis of sequenced bacterial genomes.
Resistome in the strain population according to sample origin: non-diabetic wounds | 3 - 6 months
  The presence of antibiotic resistance genes (resistome) will be identified by bioinformatics analysis of sequenced bacterial genomes.
Resistome in the strain population according to sample origin: diabetic wounds | 3 - 6 months
  The presence of antibiotic resistance genes (resistome) will be identified by bioinformatics analysis of sequenced bacterial genomes.
Resistome in the strain population according to sample origin: blood cultures | 3 - 6 months
  The presence of antibiotic resistance genes (resistome) will be identified by bioinformatics analysis of sequenced bacterial genomes.
Resistome in the strain population according to sample origin: nasal carriage | 3 - 6 months
  The presence of antibiotic resistance genes (resistome) will be identified by bioinformatics analysis of sequenced bacterial genomes.
Virulome in the strain population according to sample origin: osteitis | 3 - 6 months
  The presence of virulence genes (virulome) will be identified by bioinformatics analysis of sequenced bacterial genomes.
Virulome in the strain population according to sample origin: non-diabetic wounds | 3 - 6 months
  The presence of virulence genes (virulome) will be identified by bioinformatics analysis of sequenced bacterial genomes.
Virulome in the strain population according to sample origin: diabetic wounds | 3 - 6 months
  The presence of virulence genes (virulome) will be identified by bioinformatics analysis of sequenced bacterial genomes.
Virulome in the strain population according to sample origin: blood cultures | 3 - 6 months
  The presence of virulence genes (virulome) will be identified by bioinformatics analysis of sequenced bacterial genomes.
Virulome in the strain population according to sample origin: nasal carriage | 3 - 6 months
  The presence of virulence genes (virulome) will be identified by bioinformatics analysis of sequenced bacterial genomes.
Plasmids inthe strain population and according to sample origin: osteitis | 3 - 6 months
  The presence of plasmids will be identified by bioinformatics analysis of sequenced bacterial genomes.
Plasmids inthe strain population and according to sample origin: non-diabetic wounds | 3 - 6 months
  The presence of plasmids will be identified by bioinformatics analysis of sequenced bacterial genomes.
Plasmids inthe strain population and according to sample origin: diabetic wounds | 3 - 6 months
  The presence of plasmids will be identified by bioinformatics analysis of sequenced bacterial genomes.
Plasmids inthe strain population and according to sample origin: blood cultures | 3 - 6 months
  The presence of plasmids will be identified by bioinformatics analysis of sequenced bacterial genomes.
Plasmids inthe strain population and according to sample origin: nasal carriage | 3 - 6 months
  The presence of plasmids will be identified by bioinformatics analysis of sequenced bacterial genomes.
Phenotypic resistance profiles in the population in a subsample of 85 strains | 6 - 14 months
  The minimum inhibitory concentration for a series of antibiotics will be recorded (antibiograms of isolates).These antibiograms will be established on newly-marketed or current molecules such as Ceftarolin, Ceftobiprol, Dalbavancin, Delafloxacin, Tedizolid and Oritavancin.
Phenotypic resistance profiles in the population and according to sample origin: osteitis | 6 - 14 months
  Minimum inhibitory concentration for a series of antibiotics (antibiograms of isolates). These antibiograms will be established on newly-marketed or current molecules such as Ceftarolin, Ceftobiprol, Dalbavancin, Delafloxacin, Tedizolid and Oritavancin.
Phenotypic resistance profiles in the population and according to sample origin: non-diabetic wounds | 6 - 14 months
  Minimum inhibitory concentration for a series of antibiotics (antibiograms of isolates). These antibiograms will be established on newly-marketed or current molecules such as Ceftarolin, Ceftobiprol, Dalbavancin, Delafloxacin, Tedizolid and Oritavancin.
Phenotypic resistance profiles in the population and according to sample origin: diabetic wounds | 6 - 14 months
  Minimum inhibitory concentration for a series of antibiotics (antibiograms of isolates). These antibiograms will be established on newly-marketed or current molecules such as Ceftarolin, Ceftobiprol, Dalbavancin, Delafloxacin, Tedizolid and Oritavancin.
Phenotypic resistance profiles in the population and according to sample origin: blood cultures | 6 - 14 months
  Minimum inhibitory concentration for a series of antibiotics (antibiograms of isolates). These antibiograms will be established on newly-marketed or current molecules such as Ceftarolin, Ceftobiprol, Dalbavancin, Delafloxacin, Tedizolid and Oritavancin.
Phenotypic resistance profiles in the population and according to sample origin: nasal carriage | 6 - 14 months
  Minimum inhibitory concentration for a series of antibiotics (antibiograms of isolates). These antibiograms will be established on newly-marketed or current molecules such as Ceftarolin, Ceftobiprol, Dalbavancin, Delafloxacin, Tedizolid and Oritavancin.
Amount of biofilm formation in the absence and presence of antibiotics in a selection (85 sub-samples) of S. pettenkoferi strains according to sample origine: osteitis | 6 - 14 months
  Biofilm formation index in the presence/absence of a series of antibiotics (antibiograms of isolates). These antibiotics will be newly-marketed or current molecules such as Ceftarolin, Ceftobiprol, Dalbavancin, Delafloxacin, Tedizolid and Oritavancin. Results recorded on a scale ranging from 0 = biofilm and 12 = no biofilm
Amount of biofilm formation in the absence and presence of antibiotics in a selection (85 sub-samples) of S. pettenkoferi strains according to sample origine: non-diabetic wounds | 6 - 14 months
  Biofilm formation index in the presence/absence of a series of antibiotics (antibiograms of isolates). These antibiotics will be newly-marketed or current molecules such as Ceftarolin, Ceftobiprol, Dalbavancin, Delafloxacin, Tedizolid and Oritavancin. Results recorded on a scale ranging from 0 = biofilm and 12 = no biofilm
Amount of biofilm formation in the absence and presence of antibiotics in a selection (85 sub-samples) of S. pettenkoferi strains according to sample origine: diabetic wounds | 6 - 14 months
  Biofilm formation index in the presence/absence of a series of antibiotics (antibiograms of isolates). These antibiotics will be newly-marketed or current molecules such as Ceftarolin, Ceftobiprol, Dalbavancin, Delafloxacin, Tedizolid and Oritavancin. Results recorded on a scale ranging from 0 = biofilm and 12 = no biofilm
Amount of biofilm formation in the absence and presence of antibiotics in a selection (85 sub-samples) of S. pettenkoferi strains according to sample origine: blood cultures | 6 - 14 months
  Biofilm formation index in the presence/absence of a series of antibiotics (antibiograms of isolates). These antibiotics will be newly-marketed or current molecules such as Ceftarolin, Ceftobiprol, Dalbavancin, Delafloxacin, Tedizolid and Oritavancin. Results recorded on a scale ranging from 0 = biofilm and 12 = no biofilm
Amount of biofilm formation in the absence and presence of antibiotics in a selection (85 sub-samples) of S. pettenkoferi strains according to sample origine: nasal carriage | 6 - 14 months
  Biofilm formation index in the presence/absence of a series of antibiotics (antibiograms of isolates). These antibiotics will be newly-marketed or current molecules such as Ceftarolin, Ceftobiprol, Dalbavancin, Delafloxacin, Tedizolid and Oritavancin. Results recorded on a scale ranging from 0 = biofilm and 12 = no biofilm
Bacterial growth rate according to sample origin in a sub-sample of 20 strains: osteitis | 6 - 14 months
  Bacterial growth curve by measuring absorbance on bacterial culture over time.
Bacterial growth rate according to sample origin in a sub-sample of 20 strains: non-diabetic wounds | 6 - 14 months
  Bacterial growth curve by measuring absorbance on bacterial culture over time.
Bacterial growth rate according to sample origin in a sub-sample of 20 strains: diabetic wounds | 6 - 14 months
  Bacterial growth curve by measuring absorbance on bacterial culture over time.
Bacterial growth rate according to sample origin in a sub-sample of 20 strains: blood cultures | 6 - 14 months
  Bacterial growth curve by measuring absorbance on bacterial culture over time.
Bacterial growth rate according to sample origin in a sub-sample of 20 strains: nasal carriage | 6 - 14 months
  Bacterial growth curve by measuring absorbance on bacterial culture over time.
Virulence profiles according to sample origin in a sub-sample of 3 strains: osteitis | 6 - 14 months
  The rate of internalisation and release of LDH (a sign of cellular toxicity of the bacterial isolate) in an in vitro osteoblast cell culture model (MC3T3-E1)
Virulence profiles according to sample origin in a sub-sample of 3 strains: intracellular bacterial multiplication of S. pettenkoferi strains from osteitis | 6 - 14 months
  The amount of intracellular bacterial multiplication will be assessed in an in vitro macrophage cell culture model (RAW 264.7).
Virulence profiles according to sample origin in a sub-sample of 3 strains: diabetic wounds | 6 - 14 months
  The rate of internalisation and release of LDH (a sign of cellular toxicity of the bacterial isolate) in an in vitro osteoblast cell culture model (MC3T3-E1)
Virulence profiles according to sample origin in a sub-sample of 3 strains: intracellular bacterial multiplication of S. pettenkoferi strains from diabetic wounds | 6 - 14 months
  The amount of intracellular bacterial multiplication will be assessed in an in vitro macrophage cell culture model (RAW 264.7).
Virulence profiles according to sample origin in a sub-sample of 3 strains: blood cultures | 6 - 14 months
  The rate of internalisation and release of LDH (a sign of cellular toxicity of the bacterial isolate) in an in vitro osteoblast cell culture model (MC3T3-E1)
Virulence profiles according to sample origin in a sub-sample of 3 strains:intracellular bacterial multiplication of S. pettenkoferi strains from blood cultures | 6 - 14 months
  The amount of intracellular bacterial multiplication will be assessed in an in vitro macrophage cell culture model (RAW 264.7).
Virulence profiles according to sample origin in a sub-sample of 3 strains: nasal carriage | 6 - 14 months
  The rate of internalisation and release of LDH (a sign of cellular toxicity of the bacterial isolate) in an in vitro osteoblast cell culture model (MC3T3-E1)
Virulence profiles according to sample origin in a sub-sample of 3 strains:intracellular bacterial multiplication of S. pettenkoferi strains from nasal carriage | 6 - 14 months
  The amount of intracellular bacterial multiplication will be assessed in an in vitro macrophage cell culture model (RAW 264.7).
Virulence profiles according to sample origin in a sub-sample of 3 strains: survival time of diabetic zebrafish immersed in S. pettenkoferi strains from osteitis | Up to 48 hours
  Survival curve at 48 hours
Virulence profiles according to sample origin in a sub-sample of 3 strains: survival time of diabetic zebrafish immersed in S. pettenkoferi strains from non-diabetic wounds | Up to 48 hours
  Survival curve at 48 hours
Virulence profiles according to sample origin in a sub-sample of 3 strains: survival time of diabetic zebrafish immersed in S. pettenkoferi strains from diabetic wounds | Up to 48 hours
  Survival curve at 48 hours
Virulence profiles according to sample origin in a sub-sample of 3 strains: survival time of diabetic zebrafish immersed in S. pettenkoferi strains from blood cultures | Up to 48 hours
  Survival curve at 48 hours
Virulence profiles according to sample origin in a sub-sample of 3 strains: survival time of diabetic zebrafish immersed in S. pettenkoferi strains from nasal carriage | Up to 48 hours
  Survival curve at 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Chloé MAGNAN, Dr., Principal Investigator — Nîmes University Hospital, FRANCE
Locations (1):
- Nîmes University Hospital, Nîmes, Gard, France